CLINICAL TRIAL: NCT01692847
Title: Examination of the Impact of Better Surveillance and Communication of Patient Deterioration on Patient Related Outcomes (VitalCare - Guardian Version 2)
Brief Title: Examination of the Impact of Better Surveillance and Communication of Patient Deterioration on Patient Related Outcomes
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: SD-05163-BBN-IGS; 12/WA/0050 (Other: Research Ethics Committee)
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Severe Sepsis; Cardiac Arrest; Respiratory Failure
Keywords: patient deterioration; rapid response teams; acute care teams; early warning scoring
MeSH Terms: conditions — Sepsis; Heart Arrest; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RRT calls prior to IGS use: Patients who triggered ACT/RRT calls prior to the installation of the IGS (Intellivue Guardian System)
- RRT calls during IGS use: Patients who triggered ACT/RRT calls after the installation of IGS. All patients on the study ward receive the same care in both groups. The only difference is the system used to collect vital signs and to inform the staff about patient deteriorations. In Group 2, the IGS (FDA approved and CE marked) is the vital signs collection and information system.

SUMMARY:
A hospitals manual method of patient monitoring will be implemented in an automated system and supported by an early patient deterioration detection for timely escalation. The purpose of this study is to assess if clinical outcomes of patients in Acute Care are significantly improved by such a system.

DETAILED DESCRIPTION:
The purpose of this study is to assess if the Philips IntelliVue Guardian Solution (IGS) with all its components can significantly improve clinical outcomes for deteriorating patients on a general medical ward prior and after referral to the hospitals' Acute Care Team (ACT). Further, to provide evidence that the Philips IGS assists to increase the efficiency of a hospital's Early Warning Scoring process (afferent and efferent arm of the escalation system).

The introduction of such an intelligent automated system offers a unique opportunity to address the breakdown in the chain of prevention by strengthening the reliability of calls-for-help to responders through a technical solution with the potential for a more timely escalation where appropriate.

In this study the hospital's Standard of Care protocol for the monitoring of vital signs (including timing, vital signs collected and escalation instructions) will be implemented in a commercially available intelligent automatic monitoring and notification system. No investigational procedures or devices are associated with this protocol.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the study units during the period of data collection

Exclusion Criteria:

* less than 24h on ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to observe a non-probability, convenience sample of patients which will consist primarily of acutely ill hospitalized adult patients (at least 18 years of age). Study participants will be recruited from all eligible patients during the enrollment period who are having vital signs monitoring performed as Standard of Care.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2012-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improvement of outcome for patients after implementing the IGS | 15 months
  Does the IGS significantly increase positive outcomes for deteriorating patients after referral to the RRT/ACT as measured by the MAELOR score

SECONDARY OUTCOMES:
Early detection of patient deterioration | 15 months
  Does the IGS detect patient deterioration earlier and therefore prevent or shorten periods of severe illness.
Daily workload for the ward's personnel | 15 months
  Does the IGS reduce the daily workload related to patient surveillance for the general ward personnel.
Level of satisfaction | 15 months
  Do Nurses and Doctors express a higher level of satisfaction with the IGS in place than with their current paper-based surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Subbe, MD, Principal Investigator — Bangor University
Locations (1):
- Ysbyty Gwynedd Hospital, Bangor, Penrhosgarnedd, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Subbe CP, Duller B, Bellomo R. Effect of an automated notification system for deteriorating ward patients on clinical outcomes. Crit Care. 2017 Mar 14;21(1):52. doi: 10.1186/s13054-017-1635-z. PMID 28288655